CLINICAL TRIAL: NCT04688125
Title: Evaluation of An Optical Measurement Algorithm Combined With Patient and Provider Input to Reduce Mask Exchanges During Initial Positive Airway Pressure Therapy
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Timothy Morgenthaler, Consultant, Mayo Clinic
Other Study IDs: 20-006272
Record Dates: First submitted 2020-12-08; First posted 2020-12-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome (OHS); Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity Hypoventilation Syndrome; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Continuous positive airway pressure and non-invasive ventilation are common treatment modalities for obstructive sleep apnea, central sleep apnea, and chronic alveolar hypoventilation from a variety of causes. Use of positive airway pressure (PAP) requires use of an interface, commonly referred to as a "mask." There are a range of mask options available, differing in configuration and sizing, including masks that fit into the nostrils (nasal pillows, NP), cover the nose (nasal masks, NM), cover both the nose and the mouth (oronasal masks, ONM), and rarely those that fit into the mouth (oral masks, OM) or over the entire face. The variety of masks, sizes, and materials result from the wide variety of facial configurations and patient preferences along with requirements to provide a good seal for varying pressure requirements. Failure to find a good match for a given patient may result in significant side effects, such as eye irritation owing to leak into the eyes, skin pressure sores, noise generation, and inadequate therapy when air leaks are extreme. Pressure sores, mask dislodgement, claustrophobic complaints, air leaks, and sore eyes occur in 20-50% of patients with OSA receiving PAP, and these effects negatively correlate with PAP compliance. Furthermore, several trials point to differences in compliance related to which types of masks are utilized. In a randomized cross-over trial, compliance was 1 hour more per night in patients using NM compared to those using ONM.1 In another, NPs were associated with fewer adverse effects and better subjective sleep quality than NMs.2 Therefore, failure to find an acceptable mask results in lower or non-compliance, and therefore treatment failure.

Currently, finding a right mask is performed either using crude templates, or via an iterative process, variably guided by experts in mask fitting. There are no standard certifications or algorithms to guide mask fitting. Given the above, it would be very desirable to find a reliable method to reduce the errors in mask fitting so that the costs, inconvenience, and suffering are all reduced.

DETAILED DESCRIPTION:
Patients will be recruited from Mayo Clinic sleep medicine practices who have completed testing and are initiating PAP therapy for obstructive sleep apnea (OSA), obesity hypoventilation syndrome (OHS), or central sleep apnea syndrome (CSA). Testing will be performed for clinical reasons on patients referred for evaluation for sleep disordered breathing. Testing is at the clinician's discretion and can be either polysomnography or home sleep apnea tests. Patients meeting inclusion and not meeting exclusion criteria will be offered the opportunity to participate in this study.

Participating patients will be randomized into one of two groups: the Active group or the Usual Care. A member of the study team register each patient to use the MaskFit AR™ mobile application to take facial measurements and generate mask recommendations. The patient will then be provided with a list recommendations and will be invited to use this list to select their mask from their durable medical equipment company. This is the differentiating part of the study, with the recommendation for a mask being decided by the patient's group assignment. The recommendation for masks may or may not be different from the one written on initial prescription. After the initial visit at the study center, all participants will also be contacted for a follow-up call and will also be asked to complete brief online surveys, one after 40 days and one after 90 days following the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Sleep testing shows an apnea-hypopnea index or respiratory event index ≥5
* Patient is PAP naïve or no PAP use within the last 10 years
* Patient's diagnosis is obstructive sleep apnea, obesity hypoventilation syndrome, or central sleep apnea syndrome
* Prescribed therapy is CPAP, A-PAP, or BPAP in a spontaneous modality
* Patient is able to provide consent
* Patient is English speaking (limited to English for device)

Exclusion Criteria:

* Prescribed therapy is BPAP ST or ASV
* Patient is not able to provide consent
* Patient is not able to speak or read English
* Nasal or facial trauma or surgery that leaves atypical facial features

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female age ≥18 years old who initiating PAP therapy for obstructive sleep apnea (OSA), obesity hypoventilation syndrome (OHS), or central sleep apnea syndrome (CSA).
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mask exhange | 90 days
  Number of patient-initiated requests for mask changes during the first 90 days of PAP use
PAP Satisfaction | 90 days
  Measured using the PAP satisfaction questionnaire. CPAP Questionnaire is a 12 item questionnaire, with items 1-6 a Likert like scale asking about various types of discomfort, and questions 7-12 using a 100 mm VAS to answer questions related to PAP and sleep satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Morgenthaler, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification, may be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available throughout the study and will continue to be analyzed on an ongoing basis after the study is completed.

REFERENCES:
- [Background] Dibra MN, Berry RB, Wagner MH. Treatment of Obstructive Sleep Apnea: Choosing the Best Interface. Sleep Med Clin. 2020 Jun;15(2):219-225. doi: 10.1016/j.jsmc.2020.02.008. PMID 32386696
- [Background] Avellan-Hietanen H, Brander P, Bachour A. Symptoms During CPAP Therapy Are the Major Reason for Contacting the Sleep Unit Between Two Routine Contacts. J Clin Sleep Med. 2019 Jan 15;15(1):47-53. doi: 10.5664/jcsm.7568. PMID 30621836
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials